CLINICAL TRIAL: NCT00052845
Title: A Phase II Study Of Estramustine, Docetaxel, And Exisulind (IND #64733) In Men With Hormone Refractory Prostate Cancer
Brief Title: Docetaxel, Estramustine, and Exisulind in Treating Patients With Metastatic Prostate Cancer That Has Not Responded to Hormone Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-90004; U10CA031946 (NIH); CALGB-90004; CDR0000258766 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2003-01-24; First posted 2003-01-27 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Estramustine; sulindac sulfone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Combined chemotherapy (Experimental): combination of 3 chemotherapy agents for hormone refractory prostate cancer
  Interventions: Drug: docetaxel; Drug: estramustine phosphate sodium; Drug: exisulind

INTERVENTIONS:
Drug: docetaxel — 70 mg/sq m IV infusion over 1 hour Day 2 of ea cycle
Drug: estramustine phosphate sodium — 280 mg PO tid Days 1-5 of ea cycle
Drug: exisulind — Two 125 mg capsules PO bid Days 1-21 of ea cycle

SUMMARY:
RATIONALE: Androgens can stimulate the growth of prostate cancer cells. Estramustine may fight prostate cancer by reducing the production of androgens. Exisulind may stop the growth of prostate cancer by stopping blood flow to the tumor. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining these therapies may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining estramustine with exisulind and docetaxel in treating patients who have metastatic prostate cancer that has not responded to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the time to objective and biochemical progression and response proportion (objective and post-therapy changes in PSA) in patients with hormone refractory metastatic prostate cancer treated with docetaxel, estramustine, and exisulind.
* Determine the toxic effects of this regimen in these patients.
* Determine the overall survival of patients treated with this regimen.

OUTLINE: Patients receive oral estramustine 3 times daily on days 1-5, docetaxel IV over 1 hour on day 2, and oral exisulind twice daily on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * Progressive systemic (metastatic) disease despite castrate levels of testosterone secondary to orchiectomy or luteinizing hormone-releasing hormone (LHRH) agonist therapy

    * Castrate levels of testosterone must be maintained
    * LHRH analog therapy should be continued
  * Failed prior standard androgen-deprivation therapy
  * Serum testosterone no greater than 50 ng/mL for patients who have not had bilateral orchiectomy
* Evidence of metastatic disease on CT scan, MRI, or bone scan (no positron-emission tomography or prostascint)
* Evidence of progressive disease after most recent prior therapy (including hormonal therapy) as defined by 1 of the following:

  * Measurable disease progression

    * More than 20% increase in the sum of the longest diameters of target lesions from the time of maximal regression or the appearance of 1 or more new lesions
  * Bone scan progression

    * Appearance of 1 or more new lesions on bone scan attributable to prostate cancer AND
    * PSA at least 5 ng/mL
  * PSA progression

    * PSA at least 5 ng/mL which has increased serially from baseline on 2 occasions (at least 1 week apart) NOTE: If the confirmatory PSA is less than screening PSA, an additional test for rising PSA is required

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* AST and ALT no greater than 1.5 times upper limit of normal (ULN)
* Bilirubin no greater than ULN

Renal

* Creatinine no greater than 1.5 times ULN

Cardiovascular

* No myocardial infarction within the past year
* No significant change in anginal pattern within the past year
* No congestive heart failure
* No New York Heart Association class II-IV heart disease
* No deep vein thrombosis within the past year

Pulmonary

* No pulmonary embolus within the past year

Other

* No clinically significant peripheral neuropathy
* No known hypersensitivity to sulindac
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior cytotoxic chemotherapy (including estramustine or suramin)
* No other concurrent chemotherapy

Endocrine therapy

* See Disease Characteristics
* At least 4 weeks since prior flutamide and megestrol
* At least 6 weeks since prior bicalutamide and nilutamide
* At least 4 weeks since prior hormonal therapy known to decrease PSA levels (including ketoconazole, aminoglutethimide, finasteride, or any systemic corticosteroid)
* Concurrent primary testicular androgen suppression therapy (e.g., with a LHRH analog) allowed
* No other concurrent hormonal therapy except:

  * Steroids for adrenal insufficiency
  * Hormones for non-disease-related conditions (e.g., insulin for diabetes)
  * Intermittent dexamethasone as an antiemetic

Radiotherapy

* At least 4 weeks since prior radiotherapy and recovered
* At least 8 weeks since prior strontium chloride Sr 89 or samarium Sm 153 lexidronam pentasodium
* No concurrent palliative radiotherapy

Surgery

* See Disease Characteristics
* At least 4 weeks since prior major surgery and recovered

Other

* At least 4 weeks since prior herbal product known to decrease PSA levels (including saw palmetto, PC-SPES)
* More than 1 week since prior sulindac
* No concurrent sulindac
* No concurrent chronic nonsteroidal anti-inflammatory drugs (including COX-2 inhibitors and salicylates such as aspirin, mesalamine, salsalate, and sulfasalazine)

  * Concurrent ibuprofen and naproxen allowed
  * Low-dose aspirin (e.g., 81 mg/day) for cardiovascular prevention allowed
* No concurrent full-dose oral or parenteral anticoagulation therapy
* Concurrent bisphosphonate therapy allowed provided therapy was initiated at least 4 weeks before study and disease has progressed despite therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2002-11; Primary Completion 2006-01 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Time to progression | 24 months from study entry

SECONDARY OUTCOMES:
Toxicity | treatment up to 3 mon post treatment
Changes in PSA | During treatment then q 3 mon until ds progression
Overall Survival | 24 months from study entry

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Dawson, MD, Study Chair — University of Maryland Greenbaum Cancer Center
Locations (80):
- United States (78):
  - Northeast Alabama Regional Medical Center, Anniston, Alabama
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Cedars-Sinai Comprehensive Cancer Center at Cedars-Sinai Medical Center, Los Angeles, California
  - Veterans Affairs Medical Center - San Diego, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Cancer Center of Georgetown University Medical Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Washington, DC, Washington D.C., District of Columbia
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Memorial Regional Hospital Comprehensive Cancer Center, Hollywood, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Palm Beach Cancer Institute, West Palm Beach, Florida
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - West Suburban Center for Cancer Care, River Forest, Illinois
  - Saint Anthony Medical Center, Rockford, Illinois
  - Fort Wayne Medical Oncology and Hematology, Incorporated, Fort Wayne, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Baptist Hospital East - Louisville, Louisville, Kentucky
  - Marlene and Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Veterans Affairs Medical Center - Baltimore, Baltimore, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Lakeland Medical Center - St. Joseph, Saint Joseph, Michigan
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Veterans Affairs Medical Center - Las Vegas, Las Vegas, Nevada
  - Norris Cotton Cancer Center at Dartmouth Medical School, Lebanon, New Hampshire
  - Cooper University Hospital, Camden, New Jersey
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Elmhurst Hospital Center, Elmhurst, New York
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Veterans Affairs Medical Center - Asheville, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - NorthEast Oncology Associates, Concord, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Cape Fear Valley Health System, Fayetteville, North Carolina
  - Lenoir Memorial Hospital Cancer Center, Kinston, North Carolina
  - FirstHealth Moore Regional Hospital, Pinehurst, North Carolina
  - New Hanover Regional Medical Center, Wilmington, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Veterans Affairs Medical Center - Fargo, Fargo, North Dakota
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Lifespan: The Miriam Hospital, Providence, Rhode Island
  - Veterans Affairs Medical Center - Dallas, Dallas, Texas
  - Simmons Cancer Center at University of Texas Southwestern Medical Center - Dalas, Dallas, Texas
  - Green Mountain Oncology Group, Bennington, Vermont
  - Vermont Cancer Center at University of Vermont, Burlington, Vermont
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - Martha Jefferson Hospital, Charlottesville, Virginia
  - Virginia Oncology Associates - Norfolk, Norfolk, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Inc., Roanoke, Virginia
  - St. Mary's Medical Center, Huntington, West Virginia
  - Ministry Medical Group - Northern Region, Rhinelander, Wisconsin
- McGill University, Montreal, Quebec, Canada
- University of Puerto Rico School of Medicine Medical Sciences Campus, San Juan, Puerto Rico, Puerto Rico

REFERENCES:
- [Result] Dawson NA, Halabi S, Ou SS, Biggs DD, Kessinger A, Vogelzang N, Clamon GH, Nanus DM, Kelly WK, Small EJ; Cancer And Leukemia Group B. A phase II study of estramustine, docetaxel, and exisulind in patients with hormone- refractory prostate cancer: results of cancer and leukemia group B trial 90004. Clin Genitourin Cancer. 2008 Sep;6(2):110-6. doi: 10.3816/CGC.2008.n.017. PMID 18824434
- [Result] Dawson NA, Halabi S, Biggs DD, et al.: A phase II study of estramustine (E), docetaxel (D) and exisulind in hormone-refractory prostate cancer (HRPC): toxicity results of CALGB 90004. [Abstract] American Society of Clinical Oncology 2005 Prostate Cancer Symposium, 17-19 February 2005, Orlando, Florida. A-289, 2005.
- [Result] Dawson NA, Halabi S, Biggs DD, et al.: A phase II Study of estramustine (E), docetaxel (D) and exisulind in hormone-refractory prostate cancer (HRPC): initial results of CALGB 90004 . [Abstract] J Clin Oncol 23 (Suppl 16): A-4649, 415s, 2005.